CLINICAL TRIAL: NCT07282366
Title: Effect of a Video-Based Intervention on Depression-Related Stigma Among Adolescents
Brief Title: Video Intervention to Reduce Depression-related Stigma Among Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Jun Ou (Other)
Responsible Party: Sponsor-Investigator, Jian-Jun Ou, Principal investigator, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LYG20220038
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Depressed adolescents - video intervention on personal stigma (Experimental)
  Interventions: Behavioral: Video-Based Psychoeducation on Personal Stigma
- Depressed adolescents - control video (Placebo Comparator)
  Interventions: Behavioral: Neutral Health Education Video
- Non-depressed adolescents - video intervention on social stigma (Experimental)
  Interventions: Behavioral: Video-Based Psychoeducation on Social Stigma (Non-Depressed Adolescents)
- Non-depressed adolescents - control video (Placebo Comparator)
  Interventions: Behavioral: Neutral Health Education Video

INTERVENTIONS:
Behavioral: Video-Based Psychoeducation on Personal Stigma — Participants in this arm are depressed adolescents (PHQ-A >9) who receive a video-based psychoeducational intervention designed to reduce personal stigma toward depression. The intervention consists of short online videos (approximately 3-5 minutes each) developed by the research team and delivered through a WeChat mini-program. The videos include animated and narrative content explaining the nature of depression, correcting common misconceptions, and promoting empathy, self-acceptance, and help-seeking attitudes. The aim is to reduce internalized stigma, improve depression literacy, and encourage professional help-seeking among adolescents with depression.
  Arms: Depressed adolescents - video intervention on personal stigma
Behavioral: Video-Based Psychoeducation on Social Stigma (Non-Depressed Adolescents) — Participants in this arm are non-depressed (PHQ-A ≤ 9) adolescents who receive a video-based psychoeducational intervention aimed at reducing social stigma toward individuals with depression. The intervention consists of short online videos (approximately 3-5 minutes each) created by the research team and delivered via a WeChat mini-program. The videos use engaging animation and real-life narratives to explain the symptoms and causes of depression, challenge negative stereotypes, and promote understanding and acceptance of people experiencing depression. The goal is to decrease prejudicial attitudes and social distance toward people with depression and to enhance mental health literacy among adolescents.
  Arms: Non-depressed adolescents - video intervention on social stigma
Behavioral: Neutral Health Education Video — Participants in this arm watch a neutral health education video that serves as a control condition. The video, approximately 3-5 minutes in length, focuses on myopia prevention and eye health and contains no content related to mental health or depression. It is matched in duration and presentation style to the experimental videos to control for exposure time and viewing experience. The control video is delivered through the same WeChat mini-program platform and viewed once under the supervision of teachers, clinicians, or guardians. This condition allows for comparison of the specific effects of the depression-related stigma reduction videos with a neutral educational video of a similar format.
  Arms: Depressed adolescents - control video; Non-depressed adolescents - control video

SUMMARY:
Depression-related stigma is a major barrier to help-seeking among adolescents with depression. In China, few interventions specifically target stigma reduction in this population. This study aims to evaluate the effectiveness of a video-based psychoeducational intervention in reducing depression-related stigma and improving help-seeking attitudes among adolescents.

Adolescents aged 8-18 years are recruited from outpatient clinics and schools and screened using the Patient Health Questionnaire-9. Participants are categorized as depressed or non-depressed and randomly assigned into intervention or control groups: depressed adolescents receive a video on personal stigma, non-depressed adolescents receive a video on social stigma, while control groups watch a neutral myopia education video. The study hypothesizes that video-based education can effectively reduce stigma and promote positive help-seeking behaviors among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 8-18 years.
* Able to understand and complete questionnaires in Chinese.
* Normal or corrected-to-normal vision and hearing.
* Have at least a primary school education level.
* Provide written informed consent from both the participant and their parent or guardian.
* For the depressed group: score > 9 on the Patient Health Questionnaire for Adolescents (PHQ-A).
* For the non-depressed group: score ≤ 9 on the PHQ-A.

Exclusion Criteria:

* Presence of severe physical illness or neurological disease (e.g., traumatic brain injury).
* Cognitive impairment, intellectual disability, or significant visual/hearing impairment that prevents participation.
* Current psychotic symptoms or severe psychiatric comorbidities.
* Active suicidal or self-harming behaviors during the study period.
* Failure to comply with study procedures or withdrawal of consent.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Depression Stigma Scale | At baseline, immediately post-intervention, and week 8
  The Depression Stigma Scale is used as the primary outcome measure for participants with a baseline PHQ-A score > 9. The Depression Stigma Scale is an 18-item self-report measure rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating greater stigma toward depression
Depression social stigma scale | At baseline, imediately post-intervention, and week 8
  The Depression Social Stigma Scale is used as the primary outcome measure for participants with a baseline PHQ-A score ≤ 9. The Depression Social Stigma Scale is an 18-item self-report questionnaire rated on a 4-point Likert scale. Total scores range from 18 to 72, with higher scores indicating greater social stigma toward depression

SECONDARY OUTCOMES:
Attitudes Toward Seeking Professional Psychological Help Scale-Short Form | At baseline, imediately post-intervention, and week 8
  The ATSPPH-SF is a 10-item self-report questionnaire scored on a Likert 4-point scale. Total scores range from 0 to 30, with higher scores indicating more positive attitudes toward seeking professional psychological help.
General Help-Seeking Questionnaire | At baseline, imediately post-intervention, and week 8
  The General Help-Seeking Questionnaire assesses intentions to seek help from different sources. Responses are rated on a 7-point Likert scale. Total scores range from 18-126, with higher scores indicating greater intention to seek help.
Depression Literacy Questionnaire | At baseline, imediately post-intervention, and week 8
  The Depression Literacy Questionnaire is a 22-item self-report measure assessing knowledge about depression. Total scores range from 0 to 22, with higher scores indicating greater depression literacy.

OTHER OUTCOMES:
Program Evaluation Questionnaire | Imediately post-intervention
  The Program Evaluation Questionnaire is a self-developed questionnaire designed to assess participants' subjective experiences with the video-based depression intervention program. The questionnaire consists of 5 items covering overall evaluation of the intervention, satisfaction, perceived effectiveness, content preference, and willingness to participate in further feedback interviews. Items 2 and 3 are rated on 5-point Likert scales assessing satisfaction and agreement, whereas the remaining items are open-ended for qualitative feedback. Higher scores indicate a more positive evaluation of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Xiangya Second Hospital, Central South University, Changsha, Hunan, China